CLINICAL TRIAL: NCT05304741
Title: Drug Screening of Patient-derived Organoids From Advanced/Recurrent/Metastatic Colorectal Cancer Culture to Personalized Therapy, an Exploratory Research
Brief Title: The Culture of Advanced/Recurrent/Metastatic Colorectal Cancer Organoids and Drug Screening
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Principal Investigator, Dongling Zou, Director of Gynecologic Oncology Department, Chongqing University Cancer Hospital
Other Study IDs: CQGOG0501
Record Dates: First submitted 2022-03-20; First posted 2022-03-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer
Keywords: Drug Screening; Advanced / Recurrent / Metastatic Colorectal Cancer; Orgnoids
MeSH Terms: conditions — Colorectal Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Colorectal cancer tissues were cut into 1-3 mm3 pieces. Two random pieces were snap frozen and stored at -80℃ for DNA isolation, two random pieces were fixed in formalin for histopathological analysis, and the remainder was processed for organoids.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to establish an organoids platform and apply them to screen drugs for advanced/recurrent/metastatic colorectal cancer patients.

DETAILED DESCRIPTION:
The study was designed as a prospective, observational clinical trial in a single center. We establish organoids derived from patients with advanced/recurrent/metastatic colorectal cancer. Organoids will be validated with a combination of Next Generation Sequencing (NGS) analysis and histopathology. Drug screening assay will be performed on organoids with the chemotherapy and targeted agents, and the sensitivity and speciality will be compared with the clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participated in the study and signed informed consent;
2. ECOG score 0~2;
3. Expected survival over 6 months;
4. The serum or urine pregnancy test must be negative within 7 days before enrollment for the women of childbearing age who should agree that contraception must be used during the trial;
5. CBC: Hb≥70g/L、WBC≥3.5×109/ L 、ANC≥1.5×109/L、PLT≥80×109/L；
6. Serum ALT≤2×UL, AST≤2×ULN; Serum creatinine≤1.5×ULN；
7. Colorectal cancer was unresectable and confirmed as adenocarcinoma by histopathology. Patients have no significant symptoms in the primary lesion (no bleeding, perforation and obstruction in the primary focus). Besides, the carcinoma is potentially resectable but the patient refuses surgery;
8. Patients can comply with the research scheme according to the judgment of the researcher.

Exclusion Criteria:

1. Activity or uncontrol severe infection;
2. Liver cirrhosis, Decompensated liver disease;
3. History of immune deficiency, including HIV positive or suffering from a congenital immunodeficiency disease;
4. Chronic renal insufficiency or renal failure;
5. Other malignancies which diagnosed within 5 years or needed to be treated;
6. Myocardial infarction, severe arrhythmia and NYHA (New York heart association)≥2 for congestive heart failure
7. Concomitant diseases are treated by drugs that impair liver or kidney function, such as tuberculosis.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients suffered from advanced/recurrent/metastatic colorectal cancer which was diagnosed as adenocarcinoma and unresectable.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | 2 years
  Progression-free survival means the duration from enrollment to disease progression or death
Overall Survival | 3 years and 5 years
  Overall survival means the duration from enrollment to death due to any cause. The last follow-up time is calculated as the death time for subjects who lost follow-up

SECONDARY OUTCOMES:
Diagnostic Indicators | 2 years
  The sensitivity and specificity of organoids derived from colorectal cancer of predicting chemotherapy response of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Dongling Zou, M.D., Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
It involves patients' informed consent and research confidentiality.

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Feng RM, Zong YN, Cao SM, Xu RH. Current cancer situation in China: good or bad news from the 2018 Global Cancer Statistics? Cancer Commun (Lond). 2019 Apr 29;39(1):22. doi: 10.1186/s40880-019-0368-6. PMID 31030667
- [Background] Xie YH, Chen YX, Fang JY. Comprehensive review of targeted therapy for colorectal cancer. Signal Transduct Target Ther. 2020 Mar 20;5(1):22. doi: 10.1038/s41392-020-0116-z. PMID 32296018
- [Background] Kim M, Mun H, Sung CO, Cho EJ, Jeon HJ, Chun SM, Jung DJ, Shin TH, Jeong GS, Kim DK, Choi EK, Jeong SY, Taylor AM, Jain S, Meyerson M, Jang SJ. Patient-derived lung cancer organoids as in vitro cancer models for therapeutic screening. Nat Commun. 2019 Sep 5;10(1):3991. doi: 10.1038/s41467-019-11867-6. PMID 31488816
- [Background] Vlachogiannis G, Hedayat S, Vatsiou A, Jamin Y, Fernandez-Mateos J, Khan K, Lampis A, Eason K, Huntingford I, Burke R, Rata M, Koh DM, Tunariu N, Collins D, Hulkki-Wilson S, Ragulan C, Spiteri I, Moorcraft SY, Chau I, Rao S, Watkins D, Fotiadis N, Bali M, Darvish-Damavandi M, Lote H, Eltahir Z, Smyth EC, Begum R, Clarke PA, Hahne JC, Dowsett M, de Bono J, Workman P, Sadanandam A, Fassan M, Sansom OJ, Eccles S, Starling N, Braconi C, Sottoriva A, Robinson SP, Cunningham D, Valeri N. Patient-derived organoids model treatment response of metastatic gastrointestinal cancers. Science. 2018 Feb 23;359(6378):920-926. doi: 10.1126/science.aao2774. PMID 29472484
- [Background] Narasimhan V, Wright JA, Churchill M, Wang T, Rosati R, Lannagan TRM, Vrbanac L, Richardson AB, Kobayashi H, Price T, Tye GXY, Marker J, Hewett PJ, Flood MP, Pereira S, Whitney GA, Michael M, Tie J, Mukherjee S, Grandori C, Heriot AG, Worthley DL, Ramsay RG, Woods SL. Medium-throughput Drug Screening of Patient-derived Organoids from Colorectal Peritoneal Metastases to Direct Personalized Therapy. Clin Cancer Res. 2020 Jul 15;26(14):3662-3670. doi: 10.1158/1078-0432.CCR-20-0073. Epub 2020 May 6. PMID 32376656